CLINICAL TRIAL: NCT02769585
Title: Efficacy of Self-hypnosis for Weight Loss in Type 2 Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Levenson, David I., M.D. (Individual)
Responsible Party: Principal Investigator, David I. Levenson, MD, PI, Levenson, David I., M.D.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2016-05-08; First posted 2016-05-11 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; Weight Reduction
Keywords: Obesity; Diabetes Mellitus, Type 2; weight reduction
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Weight Loss | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-hypnosis (Experimental): Subjects underwent two group sessions one week apart with a certified hypnotherapist to teach them the process of self-hypnosis for the purpose of attaining weight loss. Subjects were asked to perform self-hypnosis once or twice a day for the duration of the one year trial.
  Interventions: Behavioral: Self-hypnosis
- CDE training (Active Comparator): Subjects underwent two group sessions one week apart with a certified diabetes educator to teach them re: diet and nutrition specifically as regards to a diabetic striving to lose weight. Subjects were asked to remain compliant with dietary restrictions for the duration of the one year trial.
  Interventions: Behavioral: CDE training

INTERVENTIONS:
Behavioral: Self-hypnosis — Self-hypnosis
  Arms: Self-hypnosis
Behavioral: CDE training — standard CDE training for an obese diabetic
  Arms: CDE training

SUMMARY:
Randomized study evaluating self-hypnosis versus certified diabetes educator training for weight loss in type 2 diabetics.

DETAILED DESCRIPTION:
Study Subjects: Approximately 74 type II diabetics will be randomized. Key inclusion criteria: overweight (BMI≥25), motivated to lose weight, and are at least 18 years of age.

Key exclusion criteria: pregnant women or women of childbearing age, currently taking medications for weight loss, enrolled in another clinical trial, or planning on having bariatric surgery. Any patient who is taking medication prescribed by a physician for depression, anxiety, or any other psychiatric disorder will be excluded. Patients on glucocorticoids in excess of Prednisone 7.5 mg or equivalent will also be excluded.

Study Design: All patients who pass screening will be administered the IPQ Test®[6]. This test stratifies patients on how they use their imagination, an important factor necessary to reach their goals. This is predictive of their potential to "persist" toward agreed upon goals. Patients will be divided into groups as follows: (Raw score 49-96 = high responders; Raw score 0-48 = Low responders).

Ultimately, subjects will be divided into four groups: The assignment of "high" versus "low" responders will be based on the results of the IPQ® test. Subjects will then be randomly assigned to intervention versus control in a 1:1 fashion. Optimally, there should be equal numbers in each group; however, the group sizes may be unequal depending on the relative proportions of high versus low responders. The four groups will be as follows:

Group I (high responders) will receive self-hypnosis using the GIFT™ (Goal Image Focusing Technique)[7] as the main means of autosuggestion and self/group motivation to lose weight.

Group II (low responders) will receive self-hypnosis (without the GIFT™ system) and self/group motivation to lose weight.

Group III (high responders) will receive standard nutrition, diet, and exercise counseling by a CDE (Certified Diabetes Educator) to serve as a control group for Group I.

Group IV (low responders) will receive standard nutrition, diet, and exercise counseling by a CDE (Certified Diabetes Educator) to serve as a control for group II.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 Diabetes
* BMI greater than 25

Exclusion Criteria:

* pregnant women of of childbearing age
* currently taking weight loss medications
* enrolled in another clinical trial
* currently taking medications for depression or anxiety
* currently taking Prednisone >7.5 mg day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in weight (BMI) | one year
  Comparison of subject's weight (BMI) from screening visit to last study visit.

SECONDARY OUTCOMES:
Waist circumference | One year
  change in waist circumference from screening visit to last study date
hemoglobin A1c | one year
  change in Hgb A1c from screening to last study visit
fasting glucose | one year
  change in fasting glucose from screening visit to last study visit
High versus low imagery | one year
  Comparison of subjects who scored high (>=48) or low (<= 47) on the IPQ questionnaire which was administered at the screening visit to all subjects. IPQ test can be found here Harte, Richard and Coller, Alan R. The Harte Coller IPQ® Inventory, Experimental Form E, New York/ The Harte Center for Hypnosis, 1986.
Compliance | one year
  Assess whether self-reported adherence with the treatment (self-hypnosis or CDE) influenced degree of weight loss
Reproducibility of IPQ | one year
  Compare results of IPQ test administered at screening with identical test administered at final study visit one year later. To assess how many subjects changed categorization between high (>=48) or low (<=47) responders. Information on IPQ can be found here: Harte, Richard and Coller, Alan R. The Harte Coller IPQ® Inventory, Experimental Form E, New York/ The Harte Center for Hypnosis, 1986.
Degree of weight loss in obese versus overweight | one year
  Determine if starting BMI influenced degree of weight loss.

CONTACTS AND LOCATIONS:
Overall Officials: David I Levenson, MD, Principal Investigator — East Coast Medical Associates

IPD SHARING:
Plan to Share IPD: Undecided
If the need arises we are happy to share data (blinded)